CLINICAL TRIAL: NCT04045067
Title: Low-voltage Areas Defragmentation in Sinus Rhythm for Radiofrequency Ablation of Persistent Atrial Fibrillation
Acronym: SCAR-AF
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Diseases; Atrial Fibrillation, Persistent
Keywords: Ablation; Low voltage areas
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: A group of patients who have pulmonary vein isolation alone, without low-voltage areas identified.
  Interventions: Procedure: Isolation of pulmonary veins
- Group 2: A group of patients who have pulmonary veins isolation alone, with low-voltage areas identified but the complementary defragmentation will not be carried out.
  Interventions: Procedure: Isolation of pulmonary veins
- Group 3: A group of patients who have pulmonary veins isolation, with low-voltage areas identified and the complementary defragmentation will be carried out.
  Interventions: Procedure: Isolation of pulmonary veins; Procedure: Ablation by radiofrequency of low-voltage areas

INTERVENTIONS:
Procedure: Isolation of pulmonary veins — Low voltage areas are identified and treated by radiofrequency. Atrial fibrillation is treated by heat produced by an electric current: radio frequency. This is an intervention that consists of blocking abnormal electrical activity, especially in the pulmonary veins.
Procedure: Ablation by radiofrequency of low-voltage areas — The defragmentation is guided by a map of fragmented potentials, made through a topography catheter, to locate the most abnormal areas that are the target of ablation.
  Groups: Group 3

SUMMARY:
This is a study evaluating the value of defragmentation of sinus rhythmic low voltage areas in addition to isolation of pulmonary veins in the removal of recurrent atrial fibrillation. The invasive procedure will be performed according to the procedures chosen by the rhythmologist and will in no way be modified by the patient's enrollment in the study. Similarly, the frequency of consultations, date and nature of the additional examinations will be defined by the physician, with the purpose of monitoring the patient.

DETAILED DESCRIPTION:
Radiofrequency ablation has become standard practice in the approach strategy for the symptomatic treatment of atrial fibrillation. The interest of substrate ablation, completing the isolation of the pulmonary veins is controversial. The usual technique for the ablation of recurrent atrial fibrillation is primarily a disconnection of the pulmonary veins, which can be accomplished by isolating the veins one by one or two by two. The isolation of the pulmonary veins is followed most often by a defragmentation of the atrium (ablation of the substrate). The defragmentation is guided by a map of fragmented potentials, made through a topography catheter, to locate the most abnormal areas that are the target of ablation. This strategy requires extensive ablation of the left atrium, with a long procedure time and repeated many radiofrequency shots. On the one hand there is a risk of complication related to the duration of intervention, but also in the longer term of occurrence of flutter scar. In addition to pulmonary vein isolation, the goal is to identify patients with sinus rhythm atrial arrhythmogenic substrate. Once the sinus rhythm has been restored by electrical cardioversion or spontaneously, a voltage map is carried out to identify the most abnormal (low voltage) areas, and intra-atrial fragmented potentials are identified, either spontaneously or spontaneously by the extra-stimulus method. Ablation of these abnormal areas may lead to better long-term results, limiting prolonged radiofrequency shots and complications associated with longer procedure times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent atrial fibrillation ablation, no specific indication restrictions or equipment used and regardless of the outcome of the procedure
* Patients participating in a biomedical research can participate in this study.

Exclusion Criteria:

* Pregnant or lactating women can not participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this protocol will be recruited by the centers that practice the procedure of ablation of persistent atrial fibrillation, by transcutaneous vein and trans-septal catheterization. Participation in this prospective observational study has been proposed to all centers practicing this procedure in France, regardless of the technique used. Inclusion in the study will be systematically offered to each patient who will benefit from this technique.
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the success rate of the procedures | month 18
  Comparison between the 3 study arms of the number of new episodes of symptomatic atrial fibrillation

SECONDARY OUTCOMES:
Evaluation of the efficiency of the procedures | Day 1
  Comparison between the 3 study arms of the duration of the intervention (in minutes), the duration of fluoroscopy (in minutes), rate of X-ray doses delivered during the procedure (in mGym² (milligray per meter²), the induction of atrial fibrillation at the end of the procedure or not.
Evaluation of the safety of the procedures | Day 1 / month 3 / month 6 / month 12 / month 18
  Comparison between the 3 study arms of the number and type of events regarding the types of procedure: pericardial effusion, pericardial drainage, vascular complication, ischemic stroke, heart failure, acute coronary syndrome, new atrial fibrillation episode, death.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEPILLIER, MD, Principal Investigator — Centre Cardiologique du Nord
Locations (9):
- France (9):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Clinique de l'Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Hôpital Privé Beauregard, Marseille
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Saint Gatien, Tours

IPD SHARING:
Plan to Share IPD: No